CLINICAL TRIAL: NCT06119386
Title: Quantum Molecular Resonance Electrotherapy in Severe Dry Eye Disease
Acronym: QMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Oculistico Borroni (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB13385-2568932022
Record Dates: First submitted 2023-10-17; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye
Keywords: Cornea; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 - Treated Eye (Experimental): Patients with treatment
  Interventions: Device: Rexon-Eye

INTERVENTIONS:
Device: Rexon-Eye — In this prospective, interventional study, 81 patients were randomly allocated to received 4 treatment sessions of QMR at one-week intervals (Rexon-Eye ® , Resono Ophthalmic, Trieste, Italy) (QRM group) or tear substitute 4 times daily, containing 0.15% sodium hyaluronate and 3% trehalose (Thealoz Duo ® , Thea Pharma, France) (SH-TH group). Outcomes measures included ocular surface disease index (OSDI) questionnaire, tear meniscus height (TMH), tear breakup time (TBUT), non-invasive breakup time (NIBUT), corneal fluorescein staining (CFS), lipid layer thickness (LLT), tear film osmolarity (OSM) and meibomian gland dysfunction (MGD) grade, which were assessed at baseline, 1-month and 3-months follow-up.

SUMMARY:
To evaluate the efficacy and safety of Quantum Molecular Resonance (QMR) treatment in patients with severe dry eye disease (DED), as well as its effects on aqueous-deficient (ADDE), evaporative (EDE) and mixed (MDE) dry eye.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of Quantum Molecular Resonance (QMR) treatment in patients with severe dry eye disease (DED), as well as its effects on aqueous-deficient (ADDE), evaporative (EDE) and mixed (MDE) dry eye.

In this prospective, interventional study, 81 patients will be randomly allocated to received 4 treatment sessions of QMR at one-week intervals (Rexon-Eye ® , Resono Ophthalmic, Trieste, Italy) (QRM group) or tear substitute 4 times daily, containing 0.15% sodium hyaluronate and 3% trehalose (Thealoz Duo ® , Thea Pharma, France) (SH-TH group).

Outcomes measures will include ocular surface disease index (OSDI) questionnaire, tear meniscus height (TMH), tear breakup time (TBUT), non-invasive breakup time (NIBUT), corneal fluorescein staining (CFS), lipid layer thickness (LLT), tear film osmolarity (OSM) and meibomian gland dysfunction (MGD) grade at baseline, 1-month and 3-months follow-up.

ELIGIBILITY:
Inclusion criteria:

-> 18 years old with a self-reported history of DED

* OSDI score ≥ 33 points
* TBUT less than 10 seconds.

Exclusion criteria:

* skin pathologies that prevent QRM treatment
* corneal infection and corneal dystrophies
* active ocular allergies
* intraocular surgery or laser ocular surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Ocular surface evaluation | 3 month
  Tear meniscus height (TMH) measured in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Oculistico Borroni, Gallarate, VA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foo VHX, Liu YC, Tho B, Tong L. Quantum molecular resonance electrotherapy (Rexon-Eye) for recalcitrant dry eye in an Asian population. Front Med (Lausanne). 2023 Sep 12;10:1209886. doi: 10.3389/fmed.2023.1209886. eCollection 2023. PMID 37771976
- [Derived] Ballesteros-Sanchez A, Sanchez-Gonzalez JM, Tedesco GR, Rocha-De-Lossada C, Russo F, Spinelli A, Ingrande I, Borroni D. Efficacy and Safety of Quantum Molecular Resonance Electrotherapy in Patients with Aqueous-Deficient, Evaporative and Mixed-Type Dry Eye: A Randomized Interventional Study. Ophthalmol Ther. 2024 Feb;13(2):495-507. doi: 10.1007/s40123-023-00868-w. Epub 2023 Dec 19. PMID 38113022